CLINICAL TRIAL: NCT04452240
Title: Clinical Study to Evaluate the Safety, Efficacy and Cost Analysis of the GORE® TAG® Conformable Thoracic Stent Graft With ACTIVE CONTROL System FOR Patients With Descending Thoracic Aortic Pathologies
Brief Title: Safety, Efficacy and Cost Analysis of the Conformable Thoracic Stent Graft With ACTIVE CONTROL
Acronym: CONFORTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Endovascular Foundation (Other)
Collaborators: W.L.Gore & Associates (Industry); Bocconi University (Other)
Responsible Party: Principal Investigator, V. Riambau, MD, PhD, Professor and chief of vascular surgery division, Endovascular Foundation
Other Study IDs: EVF01
Record Dates: First submitted 2020-06-08; First posted 2020-06-30 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Thoracic Aorta; Thoracic Aorta Aneurysm; Thoracic Aorta Abnormality
Keywords: thoracic endograft; direct cost; safety; efficacy
MeSH Terms: conditions — Aortic Aneurysm, Thoracic | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: thoracic endovascular repair — Repair of thoracic aorta lesions with the application of a dedicatet stent-graft by endovascular way.
  Other Names: TEVAR

SUMMARY:
Study Design This is a prospective, multicenter, non-randomized clinical study in patients presenting thoracic aortic pathologies.

Following a baseline assessment, the implantation procedure will be performed according to the Instructions for Use and local routine practice. A follow-up visit will be performed 30 days, 6, 12,24 and 36 months after the implantation procedure.

The investigator will perform assessments of the implantation procedure and device system and document adverse events (AE) and device deficiencies. Resources utilization and unit costs will be collected at index procedure and during follow-up. HRQoL is going to be investigated in this prospective study using the generic questionnaire EQ5D 5 levels, comparing pre- and postoperative scores.

Study Objective The objective of the study is to evaluate the safety, performance and resource utilization associated with the use of GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL systems in humans having thoracic aortic pathologies. Safety will be evaluated considering mortality and morbidity variables (mainly focused on device related complications). Efficacy will be evaluated according to the variables related to the technical and clinical successes. In addition, resource utilization and associated costs will be collected prospectively with the objective to analyze differences in resource utilization between outcome groups, landing zone groups, disease severity groups, adverse event groups and case-mix groups. We will calculate the average marginal costs increase for complications when they occurred during TEVAR or surgical revascularization (e.g., paralysis, stroke, nerve injury, lymph damages, myocardial infarction, major bleeding event, respiratory complication). Resource utilization analysis is not going to be limited to the index procedure but will continue during follow-up.

Subject Population: Elective and Urgent Thoracic aorta pathologies such as aneurysms, pseudoaneurysms, dissections, blunt thoracic aorta injury, penetrating ulcers and intramural hematoma.

Planned number of patients: A total of 200 patients. Approx. 20 study centers in 2 European countries (15 in Italy and 5 in Spain) . A subgroup of 8centers will be selected for the micro-costing analysis (7 in Italy and one in Barcelona) Expected Time to Complete Enrollment: end of 2021 (18 months).

DETAILED DESCRIPTION:
Brief Summary: Study Design This is a prospective, multicenter, non-randomized clinical study in patients presenting thoracic aortic pathologies.

Following a baseline assessment, the implantation procedure will be performed according to the Instructions for Use and local routine practice. A follow-up visit will be performed 30 days, 6, 12,24 and 36 months after the implantation procedure.

The investigator will perform assessments of the implantation procedure and device system and document adverse events (AE) and device deficiencies. Resources utilization and unit costs will be collected at index procedure and during follow-up. HRQoL is going to be investigated in this prospective study using the generic questionnaire EQ5D 5 levels, comparing pre- and postoperative scores.

Study Objective The objective of the study is to evaluate the safety, performance and resource utilization associated with the use of GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL systems in humans having thoracic aortic pathologies. Safety will be evaluated considering mortality and morbidity variables (mainly focused on device related complications). Efficacy will be evaluated according to the variables related to the technical and clinical successes. In addition, resource utilization and associated costs will be collected prospectively with the objective to analyze differences in resource utilization between outcome groups, landing zone groups, disease severity groups, adverse event groups and case-mix groups. The investigators will calculate the average marginal costs increase for complications when they occurred during TEVAR or surgical revascularization (e.g., paralysis, stroke, nerve injury, lymph damages, myocardial infarction, major bleeding event, respiratory complication). Resource utilization analysis is not going to be limited to the index procedure but will continue during follow-up.

Subject Population: Elective and Urgent Thoracic aorta pathologies such as aneurysms, pseudoaneurysms, dissections, blunt thoracic aorta injury, penetrating ulcers and intramural hematoma.

Planned number of patients: A total of 200 patients. Approx. 20 study centers in 2 European countries (15 in Italy and 5 in Spain) . A subgroup of 8centers will be selected for the micro-costing analysis (7 in Italy and one in Barcelona) Expected Time to Complete Enrollment: end of 2021 (18 months).

Detailed Description: 1. Introduction 1.1. Disease1 A thoracic aortic aneurysm (TAA) and pseudoaneurysm Type B aortic dissection (TBAD) Intramural hematoma (IMH). IMH may be a precursor to both classic AD and penetrating aortic ulcer (PAU).

Blunt thoracic aortic injury (BTAI) 1.3. Study Device Description GORE® TAG® Conformable Thoracic Stent Graft with ACTIVE CONTROL System is a device designed for the endovascular repair of TAAs, BTAIs, and TBADs of the thoracic aorta. The controlled deployment is designed to optimize accuracy, angulation, and apposition. Its conformability with enhanced control allows for optimized wall apposition even in the complex aortic anatomy 2. Study Objectives 2.1. Primary Objective(s) The primary objective of CONFORTA Clinical study is to evaluate the safety, efficacy of the GORE® TAG® Conformable Thoracic Stent Graft for the treatment of patients with Thoracic Aortic pathologies.

2.2. Secondary Objective(s) 2.2.1. Health Economic Data healthcare organizations must identify and address waste in healthcare and reduce the total cost of care. The secondary objective of this trial is focusing on patient-based costing (PBC).

To provide patient care cost a micro-costing analysis (a cost estimation method that involves the direct enumeration and costing out of every input consumed in the treatment of a particular patient) will be conducted together with an assessment of patient QoL alongside the study data collection.

2.2.2. Quality of Life data This health status information is collected before and after a procedure and provides an indication of the outcomes or quality of care delivered to the patient. Among different PROMs, the preference-based measure, such as the EQ-5D and Health Utilities Index, describes patients' responses to questions not to provide a score 3. Study Design 3.1. Description of Study Design This study is a prospective, multicenter, non-randomized single-arm study to evaluate the safety and efficacy of the GORE TAG Conformable Thoracic Stent Graft with ACTIVE CONTROL system for the treatment of patients descending Thoracic Aortic pathologies.

Centers from Italy and Spain will be invited to participate to the study. A minimum of 20 Clinical Sites (15 in Italy and 5 in Spain) will participate in this study with two hundred patients estimated in this study.

Patients may be enrolled into the study provided all inclusion and no exclusion criteria are met as specified in Section 4. Subjects will be evaluated through hospital discharge and return for follow-up visits at 30 days, 6, 12, 24 and 36 months after the implantation procedure. The cost analysis is limited to the 7 Italian centers located in Region Lombardia and one in Barcelona (Hospital Clinic of Barcelona).

3.2. Study Endpoints 3.2.1. Primary Endpoints

* Freedom from descending thoracic aorta-related mortality
* Delivery /deployment success of the study device systems

This evaluation will include the following:

* evaluation of the delivery system
* overall rate of vascular access complications (≤30 days)
* rate of access failures
* rate of deployment system difficulties
* Rate of angulation tool usage
* Rate of arterial pressure reduction maneuver 3.2.2. Secondary study endpoints
* Micro-costing analysis
* Change in QoL from baseline 4. Study Population 4.1. Description of Population Patients with Elective and Urgent Thoracic aorta pathologies such as TAAs, pseudoaneurysms, TBADs, BTAIs, PAUs and IMHs, are eligible for screening for participation in the study.

Only patients who meet all of the Inclusion Criteria and none of the Exclusion Criteria will be enrolled.

4.2. Inclusion Criteria Described in another section 4.3. Exclusion criteria: Described in another section 5. Study Procedures/Evaluations Sites are required to use a CTA scan or MRI alternatively ultrasound to assess the inserted device, permeability and integrity. Each Site will be responsible for maintaining and calibrating the equipment used.

5.1. Schedule of Events 5.2. Informed Consent Process All patients must provide informed consent prior to any study related procedures being performed. The case history (i.e., source documents/Subject chart) for each Subject shall document that such informed consent was obtained. The Ethical Committee (EC) approved consent form will be signed and personally dated by the Subject and the person who conducted the informed consent discussion. The original signed informed consent form will be retained in the Subject records. A copy of the informed consent document will be given to the Subject for their records.

5.3. Baseline Prior to entry into this study, all patients will be screened for eligibility. Screening assessments may be performed over several days and to the day of implant. The following examinations will be performed and respective data recorded 5.4. Procedure The endovascular placement of the stent-graft will be performed as described in the Instructions for Use (contains details about techniques and methods for device deployment and implantation) and according to local practice at the site.

5.5. Hospital discharge

The patients will be discharged from the clinic at the discretion of the investigator after performance of the following assessments:

* Physical examination
* Documentation of duration of intensive care unit (ICU) admission
* The investigator will document all AE and relevant concomitant medication/procedures
* Resource consumption questionnaire 5.6. Follow-Up Subjects will be evaluated through hospital discharge and return for follow-up visits at 30 days, 6, 12, 24 and 36 months after the implantation procedure.

5.7. Subject Withdrawal from the Study A Subject may withdraw from the study at any time and should notify the Investigator in this event. The Investigator may also withdraw the Subject from the study at any time based on his / her medical judgment.

5.8. Subject Lost to Follow-Up A Subject will be considered lost to follow-up and withdrawn from the study once they have missed two consecutive follow-up visits and three documented attempts have been made by the Investigator or designee to contact the Subject or next of kin.

5.9. Subject Study Completion A Subject has completed the study when final completion of all follow up visits are done. Any Subject that does not complete these requirements due to voluntary withdrawal, physician withdrawal, death, or any other reason will be considered a withdrawal..

6. Study Administration 6.1. Monitoring Site monitoring for this study will be provided by CRO Leon Research S.L.

6.2. Core Lab Core Lab services for this study will be provided by external independent observers provided by Endovascular Foundation. Core Lab assessment could be for all imaging morphometries related to 100% of the included cases or for a random sample, depending on the promoter final decision.

6.3. Protocol Deviations A Protocol deviation is defined as any change, divergence, or departure from the study design or procedures of a research protocol. The Investigator is responsible for promptly recording and reporting Protocol Deviations to the local Ethical Committee.

6.4. Protocol Amendments The Investigator will obtain EC approval on all amendments in a timely manner.

6.5. Access to Source Data/Documents Source data are defined as all information necessary for the reconstruction and evaluation of the Clinical Investigation.

The Investigator will keep all study records, source data available for inspection by the CRO's monitors, EC and regulatory authorities.

6.6. Study Records Retention The Investigator will maintain complete, accurate and current study records as required by applicable regulatory requirements. Records will be maintained during the study and for a minimum of 5 years.

6.7. Publication Plan It is the intent of the Promoter that the multicenter results of this study will be submitted for publication (in a peer reviewed journal). A publications committee will be established to review the multicenter results and develop publications at the completion of the study.

7. Data Collection and Submission 7.1. Data Collection Methods The electronic data capture system (EDC system) for this study will be provided by Xolomon Tree S.L.

7.2. Data Clarification and Correction by electronic queries 7.3. Case Report Form (CRF) Completion Schedule: 7.3.1. Baseline Demographics, clinical status and anatomical morphometrics should be provide to the data base manager prior to the inclusion and prior to the procedure 7.3.2. Procedural data should be provided with an acceptable window of 1 week after the index procedure 7.3.3. Follow-up data, Clinical and imaging information, at 1, 6, 12 and 24 months will have an acceptable window of 14 days for 1 month and 30 days for the rest.

7.3.4. Resource utilization information will be included in the CRF in combination with dedicated OR CRF 8. Risk Assessment The warnings and precautions when using the investigational device are described in detail in the Instructions for Use.

8.1. Risk-to-Benefit Rationale Risks are inherent to the endovascular repair of the thoracic aorta. Benefits are related to the repair of the pathological entity. Risk / benefit should be assessed by the physician in charge, explained to the patient and accepted, by signed informed consent, by the patient or other legal representative.

9. Adverse Events (AE) and Safety Monitoring 9.1. Anticipated AE Anticipated AE are complications that are known to be associated with thoracic aortic pathologies which are planned to undergo TEVAR with a stent-graft. See Section 8, Risk Assessment.

9.2. Unanticipated Serious Adverse Device Effects (USADE) Serious adverse device effect which by its nature, incidence, severity or outcome has not been identified in the current version of the risk analysis report. NOTE: Anticipated: an effect which by its nature, incidence, severity or outcome has been previously identified in the risk analysis report.

10. Statistical Analysis 10.1. Study Hypotheses The used thoracic endograft device, C-TAG active control, has high safety and effectiveness, in terms of very low rates of device-related complications, high accuracy on deployment and solution of the underlying pathology.

10.2. Sample Size Assumptions A cohort of a minimum of 200 cases is enough to prove our hypothesis according to previous clinical reports with similar devices. Technical improvements will be easily assessed by experienced operators with large expertise with similar devices.

10.3. Sample Size Determination That is a case series study. 200 cases are comparable with similar series already published in the literature with other similar devices for similar indications.

10.4. Data Analysis 10.4.1. Timing of Analyses An interim clinical analysis can be considered when the sample will reach 50% of the final goal.

10.4.2. Analysis Populations Consecutive patients with thoracic aorta pathology according to the inclusion and exclusion criteria previously described. The investigators will replace missing or removed cases in order to have the goal population included.

10.4.3. Statistical Analysis of Primary Endpoint(s) Quantitative parameters will be described using the following summary descriptive statistics: number of non-missing values, mean, standard deviation, median, first and third quartiles, and minimum and maximum values.

10.4.4. Statistical Analysis of Secondary Endpoint(s) The rate of MAEs will be assessed at 1 year and following time points and will be derived as: all-cause death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and secondary endovascular procedure as defined in section 9, stroke, and procedural blood loss ≥1,000mL.

11. Cost and QoL analysis 11.1. Micro-costing analysis Micro-costing analysis will be conducted to assess cost associated to each patient enrolled in the trial from the beginning of the hospitalization to the study follow-up in the perspective of the provider that need to consider budget constraints.

ELIGIBILITY:
Inclusion Criteria:

1. Male / female
2. Age between 18 and 90 years of age
3. Patient diagnosed with thoracic aorta pathology (TAA, TBAD, BTAI, PAU, IMH) suitable for TEVAR with a C-TAG Active Control stent-graft; diagnosis must be confirmed by contrast computed tomography angiography (CTA) or magnetic resonance imaging (MRI) within 3 months of the planned implant procedure.
4. Proximal and distal aortic necks suitable for stent-graft placement (i.e., inner diameter ranging between 16 and 42 mm)
5. Proximal and distal landing zones suitable for the stent-graft
6. Adequate vascular access for insertion of the delivery system
7. Written informed consent upon enrolment

Exclusion Criteria:

1. Aneurysm/lesion location not accessible to the delivery system and stent placement
2. Arterial access size insufficient for delivery system entrance or impossibility to perform a surgical access conduit
3. Treatment of lesion that would require a delivery system with usable length greater than 90 cm
4. Excessive arterial disease precluding delivery system entrance or passage
5. Systemic infection
6. Arterial tortuosity not allowing passage of the delivery system
7. Arterial or aneurysm/lesion size incompatible with stent graft
8. Mycotic aneurysm/lesions
9. Massive thrombus
10. Bleeding diathesis
11. Any condition (medical or anatomic) which makes the patient not suitable for endovascular repair according to the opinion of the investigator
12. Untreatable allergy or history of allergic reaction to radiographic contrast medium
13. Untreatable allergy or history of allergic reaction to anticoagulants
14. Hypersensitivity to any of the components of the C-TAG device
15. Participation in an investigational clinical study involving a new chemical entity or medical device within 3 months or 1 year, respectively, prior to the planned procedure
16. Patient not willing to give consent for transmission of personal "pseudonymised" data
17. For females: pregnancy or lactation
18. Women of childbearing potential (not postmenopausal or surgically sterile) not willing to use an effective method of contraception during the study. Effective methods are hormonal contraceptives (e.g., oral, implanted, or injected), intrauterine device (IUDs), and sexual abstinence.
19. Patient committed to an institution by virtue of an order issued either by the courts or by an authority
20. Patient who is unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Elective and Urgent Thoracic aorta pathologies such as TAAs, pseudoaneurysms, TBADs, BTAIs, PAUs and IMHs, are eligible for screening for participation in the study.
  Only patients who meet all of the Inclusion Criteria and none of the Exclusion Criteria will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
• Freedom from descending thoracic aorta-related mortality | 0-3 years
  Mortality rate related to the descending thoracic aorta condition or its endovascular repair or procedure
• Delivery and deployment success evaluation | during the index procedure
  it includes the following qualitative variables:
  * Delivery system evaluation
  * Overall rate of vascular access complications (≤30 days)
  * Rate of access failures
  * Rate of deployment system difficulties or failures
  * Rate of angulation tool usage
  * Rate of arterial pressure reduction maneuver

SECONDARY OUTCOMES:
o Micro-costing analysis | 0-3 years
  direct cost assessment of the total related resources to the index procedure and during the follow-up
o Change in Health-Related Quality of Life (HRQoL) as assessed using the EuroQoL Group EQ-5D (EQ-5D-5L) | 0-3 years
  assessment of the variations of the qualitty of life levels (EQ-5D-5L) pre and post procedure and during th total follow -up. There are 5 questions and 5 qualitative answers plus a numerical scale (from 0 to 100) related with the general health status.
  Numerical scale can be compared at any time of the study. Besides that, we will attribute a numerical value to the 5 qualitative answers (100 for the best/ 75, 50, 25 and 0 for the worse), and then will calculate the differences among different times during the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIAMBAU, MD. PhD, Principal Investigator — Endovascular Foundation
Locations (3):
- Italy (2):
  - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Spedali Civili di Brescia, Brescia
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Source data are defined as all information necessary for the reconstruction and evaluation of the Clinical Investigation.
  The Investigator will keep all study records, source data available for inspection by the CRO's monitors, EC and regulatory authorities.
  6.6. Study Records Retention The Investigator will maintain complete, accurate and current study records as required by applicable regulatory requirements. Records will be maintained during the study and for a minimum of 5 years.
  6.7. Publication Plan 6.7.1. It is the intent of the Promoter that the multicenter results of this study will be submitted for publication (in a peer reviewed journal). A publications committee will be established to review the multicenter results and develop publications at the completion of the study.